CLINICAL TRIAL: NCT00075608
Title: Phase II Trial of Second Autologous Transplantation in AL Amyloidosis
Brief Title: 2nd Autologous Stem Cell Transplant in Patients With Persistent/Recurrent (AL) Amyloidosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Karen Quillen, Medical Director, Blood Bank, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000347379; H-22603 (Other: Boston University Medical Center IRB)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2nd Stem Cell Transplant (Experimental): Mobilization with filgrastim autologous stem cell transplantation with melphalan conditioning stem cell infusion
  Interventions: Biological: filgrastim; Drug: melphalan; Procedure: autologous stem cell transplantation; Procedure: stem cell infusion

INTERVENTIONS:
Biological: filgrastim — 16mcg/kg IV daily beginning three days prior to stem cell collection through last day of stem cell collection
  Other Names: G-CSF
Drug: melphalan — 140-200 mcg/kg IV over two days
  Other Names: alkeran
Procedure: autologous stem cell transplantation — infusion of previously collected stem cells on Day 0
Procedure: stem cell infusion — infusion of previously collected stem cells on Day 0

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of plasma cells, either by killing the cells or by stopping them from dividing. Having a stem cell transplant to replace the blood-forming cells destroyed by chemotherapy, allows higher doses of chemotherapy to be given so that more plasma cells are killed. By reducing the number of plasma cells, the disease may progress more slowly.

PURPOSE: This phase II trial is studying how well autologous stem cell transplant works in treating patients with persistent or recurrent primary systemic (AL) amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and tolerability of second autologous stem cell transplantation in patients with persistent or recurrent AL amyloidosis.
* Determine the response rate and durability of response in patients treated with this regimen.
* Determine immune reconstitution in patients treated with this regimen.

OUTLINE:

* Mobilization: Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning before the initiation of stem cell collection and continuing until the day before the completion of stem cell collection.
* Preparative regimen: Patients receive high-dose melphalan IV over 20 minutes on days -3 and -2.
* Autologous stem cell transplantation: Autologous stem cells are reinfused on day 0.

Patients are followed at 6 months, 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 19 patients will be accrued for this study within 5-6 years.

ELIGIBILITY:
Inclusion criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed AL amyloidosis

  * Persistent or recurrent disease after 1 course of prior high-dose chemotherapy
* Previously treated with autologous stem cell transplantation
* Significant initial improvement in organ function after prior high-dose melphalan, defined by at least 1 of the following:

  * Complete hematologic remission (e.g., absence of monoclonal spike by immunofixation in serum and urine AND less then 5% plasma cells in bone marrow with no clonal predominance) OR partial hematologic response (e.g., any decrease in serum or urine monoclonal protein OR decrease in bone marrow plasmacytosis)
  * Greater than 50% reduction in proteinuria with preservation of creatinine clearance
  * Greater than 50% reduction in alkaline phosphatase OR at least 2 cm decrease in liver size by physical exam
  * Subjective neurologic improvement, as confirmed by neurologist
  * Cardiac stabilization of disease confirmed by echocardiography defined as less than 2 mm increase in mean wall thickness and/or less than 20 g increase in left ventricular mass
  * Improvement in performance status* NOTE: *This criteria alone does not constitute significant improvement in organ function
* Prior stem cell yield must have been ≥ 2 x 10^6 CD34+ cells/kg

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics
* No chemotherapy after first transplantation

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* Southwest Oncology Group- 0-2

Life expectancy

* More than 6 months

Hematopoietic

* See Disease Characteristics

Hepatic

* See Disease Characteristics

Renal

* See Disease Characteristics

Cardiovascular

* See Disease Characteristics
* Left ventricular ejection fraction ≥ 45% by multiple gated acquisition scan or echocardiogram

Pulmonary

* diffusing capacity of lung for carbon monoxide ≥ 50%

Exclusion Criteria:

* No myelodysplastic syndromes
* No abnormal bone marrow cytogenetics

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Acceptable toxicity from first transplantation, confirmed by the transplant team
* HIV negative
* No other concurrent malignancy except treated skin cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Quillen, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from March 2003 through July 2008 through the transplant clinic and amyloid clinic.
Groups:
- Second Transplant: Participants underwent a second treatment with high dose chemotherapy and stem cell transplant
Period: Overall Study
Arm/Group | Second Transplant
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Second Transplant
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.25 (1)
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Tolerability
Description: Feasibility and tolerability will be evaluated based on participants completing second transplant with tolerable adverse events
Time Frame: 3 months after treatment and annually
Population: No data were collected or analyzed due to study termination
Arm/Group | Second Transplant
Number analyzed (Participants) | 0

2. Primary Outcome: Response and Durability of Response
Description: Response and durability of response will be based on hematologic Complete Response or Partial Response and date of relapse or death
Time Frame: 3 months after treatment and annually
Population: No data were collected or analyzed due to study termination
Groups:
- 2nd SCT: Mobilization with filgrastim Second autologous peripheral blood stem cell transplant with melphalan conditioning
  filgrastim: 16mcg/kg IV daily beginning three days prior to stem cell collection through last day of SCC
  melphalan: 140-200 mcg/kg IV over two days
  autologous bone marrow transplantation: infusion of previously collected stem cells on Day 0
  peripheral blood stem cell transplantation: infusion of previously collected stem cells on Day 0
Arm/Group | 2nd SCT
Number analyzed (Participants) | 0

3. Primary Outcome: Evaluate Immune Reconstitution
Description: Evaluate immune reconstitution based on time to engraftment
Time Frame: 3 months after treatment and annually
Population: No data were collected or analyzed due to study termination
Groups:
- 2nd SCT: Mobilization with filgrastim Second autologous peripheral blood stem cell transplant with melphalan conditioning
  filgrastim: 16mcg/kg IV daily beginning three days prior to SCC through last day of SCC
  melphalan: 140-200 mcg/kg IV over two days
  autologous bone marrow transplantation: infusion of previously collected stem cells on Day 0
  peripheral blood stem cell transplantation: infusion of previously collected stem cells on Day 0
Arm/Group | 2nd SCT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were assessed for up to 1 year.
Groups:
- Second Transplant: Participants who received a second transplant
Arm/Group | Second Transplant
Serious Adverse Events (participants affected / at risk) | 12/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Second Transplant (N=12)
Sepsis (Blood and lymphatic system disorders) | 2 (3) — Grade IV
febrile neutropenia (Infections and infestations) | 8 (8) — Grade III and IV
Acute renal failure (Renal and urinary disorders) | 2 (2) — Grade IV
fatigue (General disorders) | 8 (8) — Grade III and IV
nausea (Gastrointestinal disorders) | 3 (3) — Grade III
diarrhea (Gastrointestinal disorders) | 5 (5) — Grade III
hypotension (Cardiac disorders) | 5 (5) — Grade III
arrhythmia (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Second Transplant (N=12)
nausea (Gastrointestinal disorders) | 9 (13)
diarrhea (Gastrointestinal disorders) | 5 (6)
peripheral edema (Blood and lymphatic system disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
hypocalcemia (Investigations) | 2 (2)
hypoalbuminemia (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes